CLINICAL TRIAL: NCT04131855
Title: The Omission of Pumice Prophylaxis on Bracket Failure Rates Using Self Etch Primers: A Randomized Controlled Clinical Trial
Brief Title: The Omission of Pumice Prophylaxis on Bracket Failure Rates Using Self Etch Primers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Kaminii A/P Thevadass, Principal Investigator, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DF CD1909/0057(P)
Record Dates: First submitted 2019-10-17; First posted 2019-10-18 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Orthodontic Appliance Complication
Keywords: self etch primers; pumice; orthodontic bracket failure

STUDY DESIGN:
Intervention Model Description: Participants will be placed in two different groups based on the randomization and will receive, or not receive the intervention, which is pumicing prior to bond-up, for the duration of the study.
Who Masked: Participant
Masking Description: The procedures, data collection and data analysis will be done by the orthodontic post-graduate student who is the main investigator in this study, and will not be blinded.The patients will be blinded. This will be done by pumicing the occlusal surfaces of the teeth that are in the study quadrant, and the labial surfaces of the teeth in the control quadrant. The trial is hence a single-blinded study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pumice prophylaxis. (Active Comparator): Will receive pumice prophylaxis in a slurry of plain pumice and water for 5 seconds per tooth using a rubber cup in a slow contra-angle handpiece. The teeth involved will then be washed and dried prior to using the self etch primer.
  Interventions: Other: Pumice prophylaxis
- No pumice prophylaxis. (Experimental): Will not receive pumice prophylaxis. Teeth will be washed and dried before using the self etch primer.
  Interventions: Other: No pumice prophylaxis

INTERVENTIONS:
Other: Pumice prophylaxis — Pumicing the teeth is the recommended prophylaxis to be used prior to the application of the self etch primer by the manufacturer - 3M Unitek Transbond Plus Self Etch Primer which will be used in the experiment.
  Other Names: Pumice slurry; Pumice powder
  Arms: Pumice prophylaxis.
Other: No pumice prophylaxis — Pumice prophylaxis will not be used as per manufacturers instructions.
  Arms: No pumice prophylaxis.

SUMMARY:
The aim of the study is to investigate the role of pumice prophylaxis in the self etch primer method on clinical bond strengths. The relevance is that removal of the pumicing step in the SEP method could potentially save time & cost for clinicians, and decrease discomfort for patients if it does not affect bond strengths.

The null hypothesis that will be tested is that pumice prophylaxis does not affect orthodontic bracket failure rates when used with the self etch primer. The alternative hypothesis is that there are less orthodontic bracket failures in the pumiced group while using the self etch primer.

DETAILED DESCRIPTION:
INTRODUCTION:

There is a clinically significant variation in individual understandings and approaches among orthodontists to pumicing prior to using the SEP to bond brackets. There is also a lack of current studies in the last decade comparing bond strengths between pumiced and non-pumiced teeth while using the latest SEP products in the market. Therefore the aim of this research is to the investigate the relevance of pumicing prior to bonding orthodontic brackets. The investigators also then aim to recommend either the continued usage of, or to highlight it's clinical redundancy in the bond-up process, hence reducing cost and saving time for both the patient and clinician.

SAMPLE SIZE CALCULATION:

Based on the expected proportions of bracket breakages in pumiced and non-pumiced groups, a one-tailed priori power calculation determined that 266 orthodontic brackets would be required to give a power of 0.9 at significance level of 0.05, assuming failure proportions of 2.46% and 11.41% (Lill, 2008), which was deemed a clinically significant difference.

Incorporating an attrition rate of 20%, the ideal sample size to achieve a statistically significant result would be 319 brackets, equivalent to 20 patients with 16 orthodontic brackets each.

RANDOMIZATION:

The block randomization technique will be used. A 1:1 ratio will be used with fixed block sizes of 4:4:4:4:4. There will be no stratification used in the randomisation. A computer generated random number list will be prepared by a supervisor with no clinical involvement in the trial. The allocation sequence will be concealed from the main investigator enrolling the participants in sequentially numbered, opaque and sealed envelopes.

To prevent subversion of the allocation sequence, the name and date of birth of the participant will be written on the envelope. Corresponding envelopes were opened only after the enrolled participants for that block completed all baseline assessments and it was time to allocate the intervention. Each participant will receive either an odd or even numbered envelope. The split mouth contra-lateral technique will be used. Patients receiving an even number will receive pumicing on the maxillary left and mandibular right quadrants, and patients receiving an odd number will receive pumicing on the maxillary right and mandibular left quadrants.

INTERVENTIONS:

Patients who attend the Faculty of Dentistry, University of Malaya requesting orthodontic treatment will be screened. Patients who fulfil the inclusion and exclusion criteria will be selected for this study. During screening, the participants will receive information leaflets and detailed explanations on the study. Informed consent will then be taken from the patients. A total of 20 participants will be recruited for the study.

The first appointment will be for bond-up.At the bond up appointment, the teeth will be isolated with a cheek retractor and a saliva ejector. In the control quadrants, the teeth are polished with a slurry of plain pumice and water for 5 seconds per tooth, using a rubber cup in a slow contra-angle handpiece. In the study quadrants, no pumicing will be performed. All quadrants will then washed with water and each tooth air-dried for 5 seconds. The single etch primer (SEP) Transbond Plus 3M will be then applied according to manufacturer's instructions. For each tooth, the applicator will be used to rub the enamel to be bonded for 3 seconds, the applicator returned to the well, and the process repeated for each tooth. Transbond XT adhesive will be applied to the bracket base, the brackets are placed on the teeth with brackets holders and firmly seated .Excess adhesive will be removed from around the periphery using a probe, and each bracket light-cured for 5 seconds per interspace with an LED curing light. (Planmeca Lumion).

The brackets used will be mesh-based stainless steel orthodontic brackets (3M Unitek Gemini MBT 0.022"x 0.028) and the wires used will be 3M Unitek Nitinol (NiTi) HANT & Stainless Steel (SS) wires. A check for occlusal interferences will be made and the initial 0.014 NiTi archwires will be placed in all four quadrants after band cementation and secured with elastomeric ligatures. Post-operative patient instructions will be given.

To maximize moisture control and standardize all patients, the teeth will be bonded in a specific order as follows: first, the upper labial segment followed by the lower labial segment, then the right premolars (uppers then lowers) and finally the left premolars(uppers then lowers).

The wire sequence used will be 0.014 Niti to 0.018 NiTi to 17x25 NiTi to 19x25 Stainless Steel archwire. Patients are required to be in the 19x25 SS wire for at least a month.

DATA COLLECTION:

Any bond failure that occurs until the patient is in the 19x25 SS wire for a month, will be verified by the clinician. The patient's name along with the position of the bracket and the amount of adhesive remnant left on the surface will be recorded in a logbook as per the Adhesive Remnant Index (ARI).

Any brackets that debond during treatment will be rebonded with Transbond XT after conventional acid-etching with 37% phosphoric acid. They will then be subsequently excluded from the trial to avoid recounts. Bond failures were recorded prospectively, as was the adhesive remnant index (ARI) results. Data on bond failure will be collected at 1 month after placement of the 19x25 SS wire.

The central and lateral incisors will be grouped as anterior teeth, and the canines and premolars will be grouped as posterior teeth for recording purposes.

STATISTICAL METHODS:

Statistical Analysis will be done using SPSS software version 22. P < 0.05 will be set as the level of significance.

The Shapiro-Wilk test of normality (n<50) will be done to determine if the data is normally distributed.

The independent T-test will then be used to compare the means of both groups, pumiced and non-pumiced to determine if there is a statistically significant difference between both the groups.

If the results are not distributed normally, the non-parametric Mann Whitney U-test will be used to compare the means.

ADDITIONAL ANALYSIS:

1. The independent T-test/ Mann-Whitney U-test will be used to compare means to assess the difference in breakage failures between the anterior and posterior groups.
2. The Levene's test of variance will be applied to the results of the Adhesive Remnant Index (ARI), if the variances are equal, the one way analysis of variance (ANOVA) test will be used to determine if there is a statistically significant differences between the means of the results. If the variances are assumed to be unequal, the Kruskal-Wallis test will be used for this purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving fixed appliance therapy with only metal brackets on both upper and lower arches.
2. Good oral hygiene.
3. Balanced extractions in both upper and lower arches.
4. Right-handed patients

Exclusion Criteria:

1. Enamel defects, hypoplasia or buccal restorations that would preclude bonding to enamel.
2. Orthognathic cases.
3. Surgically exposed teeth or teeth where bracket placement will be delayed.
4. Patients with craniofacial anomalies.
5. Previous use of fixed appliances.
6. Patients that will require partial ligation of teeth immediately after bond-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-02-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
To compare the bond failure rates between pumiced and non-pumiced teeth. | Data on bond failure will be collected at 1 month after placement of the 19x25 SS wire.
  Done by calculating and comparing the percentage of bracket breakages between the pumiced and non-pumiced quadrants.

SECONDARY OUTCOMES:
To compare the bracket breakage rates between anterior and posterior teeth. | Data on bond failure will be collected at 1 month after placement of the 19x25 SS wire.
  Done by calculating and comparing the percentage of bracket breakages in anterior and posterior teeth in both the groups.
To determine the interfaces at which the bond failures occur after bracket breakage. | Data on adhesive remnant will be collected from the tooth surface immediately after bracket breakage.
  Done by assessing the amount of adhesive remnant remaining on the tooth surface.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kaminii Thevadass, BDS, Principal Investigator — Department of Paediatric Dentistry and Orthodontics,University of Malaya.; Prof Dr Siti Adibah Othman, BDS, Study Director — Department of Paediatric Dentistry and Orthodontics,University of Malaya.; Dr Nor Nadia Zakaria, BDS, Study Director — Department of Paediatric Dentistry and Orthodontics,University of Malaya.

IPD SHARING:
Plan to Share IPD: No
Consent has not yet been gained from participants as recruiting has not begun.

REFERENCES:
- [Result] Burgess AM, Sherriff M, Ireland AJ. Self-etching primers: is prophylactic pumicing necessary? A randomized clinical trial. Angle Orthod. 2006 Jan;76(1):114-8. doi: 10.1043/0003-3219(2006)076[0114:SPIPPN]2.0.CO;2. PMID 16448279
- [Result] Lill DJ, Lindauer SJ, Tufekci E, Shroff B. Importance of pumice prophylaxis for bonding with self-etch primer. Am J Orthod Dentofacial Orthop. 2008 Mar;133(3):423-6; quiz 476.e2. doi: 10.1016/j.ajodo.2006.03.039. PMID 18331943